CLINICAL TRIAL: NCT02801825
Title: A Randomized Study of Ultrasound-guided Axillary and Femoral Artery Cannulation in Mechanically Ventilated Critically Ill Patients.
Brief Title: Ultrasound-guided Axillary Artery vs Femoral Artery Cannulation.
Acronym: AxFemArt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniwersytecki Szpital Kliniczny w Opolu (Other)
Responsible Party: Principal Investigator, Ryszard Gawda, MD PhD, Ryszard Gawda, MD PhD, Uniwersytecki Szpital Kliniczny w Opolu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AxFemArt
Record Dates: First submitted 2016-06-07; First posted 2016-06-16 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Critical Illness
Keywords: axillay artery; cannulation; femoral artery
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Axillary artery. (Experimental): Cannulation of the axillary artery.
  Interventions: Procedure: Real-time ultrasound-guided in-plane infraclavicular axillary artery cannulation.
- Femoral artery. (Experimental): Cannulation of the femoral artery.
  Interventions: Procedure: Real-time ultrasound-guided out-of-plane femoral artery cannulation.

INTERVENTIONS:
Procedure: Real-time ultrasound-guided in-plane infraclavicular axillary artery cannulation. — Real-time ultrasound-guided in-plane infraclavicular axillary artery cannulation.
  Arms: Axillary artery.
Procedure: Real-time ultrasound-guided out-of-plane femoral artery cannulation. — Real-time ultrasound-guided out-of-plane femoral artery cannulation.
  Arms: Femoral artery.

SUMMARY:
The main purpose of the study is to compare two ultrasound-guided arterial cannulation procedures: in-plane infraclavicular axillary artery cannulation and out-of-plane femoral artery cannulation.

ELIGIBILITY:
Inclusion Criteria:

mechanically ventilated critically ill patients with indications for artery cannulation:

* in whom radial artery cannulation is unable to perform or
* in order to conduct hemodynamic monitoring using transpulmonary thermodilution

Exclusion Criteria:

* age less than 18 years
* trauma and hematoma at the catheterization site
* clinically significant coagulation disorders
* infection at the catheterization site
* lack of patients or closest relatives contents
* precedent surgery operation into the femoral and axillary arteries
* clinically significant ischemia of the limb at the cannulation side

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Cannulation success rate | 24 hours
  The goal of the assessment of the cannulation success rate is essential for the estimation of the usefulness of both artery approaches in clinical practice.

SECONDARY OUTCOMES:
Procedure complication rate. | 24 hours
  The goal of the assessment of the early mechanical complication rate is crucial for the estimation of the safety of both procedures in clinical practice.
Number of puncture attempts. | 24 hours
  The goal of the assessment is the evaluation which approach is easier to perform.

CONTACTS AND LOCATIONS:
Overall Officials: Ryszard Gawda, MD PhD, Principal Investigator — Department of Anesthesiology and Intensive Care, Uniwersytecki Szpital Kliniczny w Opolu
Locations (1):
- Department of Anesthesiology and Intensive Care, Uniwersytecki Szpital Kliniczny w Opolu, Opole, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gawda R, Marszalski M, Piwoda M, Molsa M, Pietka M, Filipiak K, Miechowicz I, Czarnik T. Infraclavicular, Ultrasound-Guided Percutaneous Approach to the Axillary Artery for Arterial Catheter Placement: A Randomized Trial. Crit Care Med. 2024 Jan 1;52(1):44-53. doi: 10.1097/CCM.0000000000006015. Epub 2023 Aug 7. PMID 37548510